CLINICAL TRIAL: NCT00815711
Title: Inflammation in Interstitial Lung Disease/Idiopathic Pulmonary Fibrosis
Brief Title: Idiopathic Pulmonary Fibrosis Registry for Future Studies
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Sponsor
Other Study IDs: 2007H0002
Record Dates: First submitted 2008-12-29; First posted 2008-12-30 (Estimated); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Lung Disease, Interstitial; Idiopathic Pulmonary Fibrosis
Keywords: IPF
MeSH Terms: conditions — Lung Diseases, Interstitial; Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood serum BAL fluid lung biopsy
Oversight: Data Monitoring Committee: No

SUMMARY:
To establish a registry of patients for future studies of Inflammation in Interstitial Lung Disease/Idiopathic Pulmonary Fibrosis.

DETAILED DESCRIPTION:
To establish a framework in which biologic samples and physiologic measures from patients with IPF can be longitudinally collected and evaluated. Having a bank of samples that are correlated with physiologic measures that follow patients through their course will allow the following proposed studies as well as future investigations to be efficiently carried out.

ELIGIBILITY:
Inclusion Criteria:

* any patient referred to the Interstitial Lund Disease clinic who is undergoing evaluation and or treatment for a new diagnosis of ILD. This can include patients referred for presumed pulmonary fibrosis/interstitial pneumonitis (IPF, UIP, NSIP), sarcoidosis, hypersensitivity pneumonitis, cryptogenic organising pneumonia, drug-induced, or other idiopathic ILDs.

Exclusion Criteria:

* pregnancy
* inability to follow study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2008-12-01 (Actual); Primary Completion 2015-06-10 (Actual); Study Completion 2015-06-10 (Actual)

PRIMARY OUTCOMES:
Framework | 7 + years
  To establish a framework in which biologic samples and physiologic measures from patients with IPF can be longitudinally collected and evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Clay B Marsh, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States